CLINICAL TRIAL: NCT01401543
Title: LY2452473 Formulation Exploratory Bioavailability Study
Brief Title: A Bioavailability Study of LY2452473 and Tadalafil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13326; I4K-MC-GPEA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Erectile Dysfunction
Keywords: testosterone; energy; libido; erectile function; weak muscles
MeSH Terms: conditions — Erectile Dysfunction | interventions — LY2452473; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5 mg LY2452473 + 5 mg Tadalafil (Active Comparator): 5-mg LY2452473 oral capsule and 5-mg tadalafil oral tablet, administered orally, once only. There will be a washout period of at least 7 days between doses of study drug.
  Interventions: Drug: LY2452473; Drug: Tadalafil
- LY900010 (particle size #1) (Experimental): Single combination tablet containing 5 mg tadalafil and 5 mg LY2452473 with a smaller particle size (d90 = 10 microns), administered orally, once only. There will be a washout period of at least 7 days between doses of study drug.
  d90 is a measurement of the distribution of particle widths such that 90% of the particles have a diameter less than the specified value.
  Interventions: Drug: LY900010
- LY900010 (particle size #2) (Experimental): Single combination tablet containing 5 mg tadalafil and 5 mg LY2452473 with an intermediate particle size (d90 = 25 microns), administered orally, once only. There will be a washout period of at least 7 days between doses of study drug.
  d90 is a measurement of the distribution of particle widths such that 90% of the particles have a diameter less than the specified value.
  Interventions: Drug: LY900010
- LY900010 (particle size #3) (Experimental): Single combination tablet containing 5 mg tadalafil and 5 mg LY2452473 with a larger particle size (d90 = 40 microns), administered orally, once only. There will be a washout period of at least 7 days between doses of study drug.
  d90 is a measurement of the distribution of particle widths such that 90% of the particles have a diameter less than the specified value.
  Interventions: Drug: LY900010

INTERVENTIONS:
Drug: LY2452473 — Administered orally
  Arms: 5 mg LY2452473 + 5 mg Tadalafil
Drug: Tadalafil — Administered orally
  Other Names: LY450190; Cialis
  Arms: 5 mg LY2452473 + 5 mg Tadalafil
Drug: LY900010 — Administered orally
  Arms: LY900010 (particle size #1); LY900010 (particle size #2); LY900010 (particle size #3)

SUMMARY:
This study compares LY2452473 taken orally as a 5 milligram (mg) capsule at the same time as a 5 mg tadalafil tablet with three different combination tablets (LY900010) of 5 mg LY2452473 and 5 mg tadalafil taken orally. The study will evaluate the amount of LY2452473 and tadalafil circulating in the blood for each treatment. Side effects will be documented. This study is approximately 34 days not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male, as determined by medical history and physical examination
* Are between a body mass index of 18.5 and 30 kilograms per meter squared (kg/m²), inclusive at screening
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Normal blood pressure and heart rate (HR; sitting) as determined by the investigator
* Have venous access sufficient to allow blood sampling
* Are reliable and willing to make themselves available for the duration of the study, and will abide by the research unit policies and procedures and study restrictions
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site
* Men must agree to use a reliable method of birth control (for example, vasectomy, condom with contraceptive foam, abstinence, or female partner's use of oral contraceptives or Norplant®; a reliable barrier method of birth control [diaphragm with contraceptive jelly]; or intrauterine device), during the study and for 1 month following the last dose of study drug

Exclusion Criteria:

* Have known allergies to LY2452473, tadalafil, or related compounds
* History of severe allergies or multiple adverse drug reactions
* Have a history or presence of cardiovascular, respiratory, hepatic (including history of cholecystectomy), renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Any abnormality in the 12-lead electrocardiogram (ECG) that in the opinion of the investigator places the subject at an unacceptable risk for study participation
* Show evidence of significant active neuropsychiatric disease
* History of significant retinal pathology
* Have a history of glaucoma
* Have a history of unexplained syncope episodes
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Show evidence of human immunodeficiency virus (HIV) and/or positive HIV antibodies
* Intended use of over-the-counter or herbal remedies within 7 days prior to dosing or during the study
* Intended use of prescription medication within 14 days prior to dosing or during the study
* Are not willing to refrain from consumption of any food, or drink any beverage containing grapefruit, pomelo, or starfruit for at least 2 weeks prior to the start of the study until its conclusion
* Heavy caffeine drinkers defined by a regular intake of more than 5 cups of coffee (or equivalent in xanthine-containing beverages) per day or subjects who have not had consistent daily caffeine consumption for 1 month prior to study entry or subjects not willing to maintain consistent caffeine consumption during the study
* Use of drugs of abuse, as evidenced by history, and/or positive findings on urinary drug screening
* Have an average weekly alcohol intake that exceeds 14 units per week or are unwilling to stop alcohol consumption for the duration of the study (1 unit = 12 ounces [oz] or 360 milliliters (mL) of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Is currently a smoker or uses tobacco products on a regular basis and has not had consistent daily tobacco use for 1 month prior to study entry or subjects not willing to maintain consistent tobacco use during the study
* Have a history of blood donation of 1 unit (approximately 450 mL) or more in the last 3 months prior to study entry
* Have previously completed or withdrawn from this study or any other study investigating LY2452473
* Within 30 days of the initial dose of study drug, have received treatment with a drug that has not received regulatory approval for any indication
* Deemed unsuitable by the investigator for any other reason
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device (other than the study drug/device used in this study), or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: First intervention: A 5-milligram (mg) LY2452473 capsule and 5-mg tadalafil tablet administered orally, once.
  Second intervention: A single combination tablet LY900010 (containing 5 mg LY2452473 with a larger particle size #3, d90 = 40 microns, and 5 mg tadalafil) administered orally, once.
  Third intervention: A single combination tablet LY900010 (containing 5 mg LY2452473 with a smaller particle size #1, d90 = 10 microns, and 5 mg tadalafil) administered orally, once.
  Fourth intervention: A single combination tablet LY900010 (containing 5 mg LY2452473 with an intermediate particle size #2, d90 = 25 microns, and 5 mg tadalafil) administered orally, once.
  There was a washout period of at least 7 days between each intervention. d90 is a measurement of the distribution of particle widths such that 90% of the particles have a diameter less than the specified value.
- Sequence 2: First intervention: A single combination tablet LY900010 (containing 5 mg LY2452473 with a smaller particle size #1, d90 = 10 microns, and 5 mg tadalafil) administered orally, once.
  Second intervention: A 5-mg LY2452473 capsule and 5-mg tadalafil tablet administered orally, once.
  Third intervention: A single combination tablet LY900010 (containing 5 mg LY2452473 with an intermediate particle size #2, d90 = 25 microns, and 5 mg tadalafil) administered orally, once.
  Fourth intervention: A single combination tablet LY900010 (containing 5 mg LY2452473 with a larger particle size #3, d90 = 40 microns, and 5 mg tadalafil) administered orally, once.
  There was a washout period of at least 7 days between each intervention. d90 is a measurement of the distribution of particle widths such that 90% of the particles have a diameter less than the specified value.
- Sequence 3: First intervention: A single combination tablet LY900010 (containing 5 mg LY2452473 with an intermediate particle size #2, d90 = 25 microns, and 5 mg tadalafil) administered orally, once.
  Second intervention: A single combination tablet LY900010 (containing 5 mg LY2452473 with a smaller particle size #1, d90 = 10 microns, and 5 mg tadalafil) administered orally, once.
  Third intervention: A single combination tablet LY900010 (containing 5 mg LY2452473 with a larger particle size #3, d90 =40 microns, and 5 mg tadalafil) administered orally, once.
  Fourth intervention: A 5-mg LY2452473 capsule and 5-mg tadalafil tablet administered orally, once.
  There was a washout period of at least 7 days between each intervention. d90 is a measurement of the distribution of particle widths such that 90% of the particles have a diameter less than the specified value.
- Sequence 4: First intervention: A single combination tablet LY900010 (containing 5 mg LY2452473 with a larger particle size #3, d90 = 40 microns, and 5 mg tadalafil) administered orally, once.
  Second intervention: A single combination tablet LY900010 (containing 5 mg LY2452473 with an intermediate particle size #2, d90 = 25 microns, and 5 mg tadalafil) administered orally, once.
  Third intervention: A 5-mg LY2452473 capsule and 5-mg tadalafil tablet administered orally, once.
  Fourth intervention: A single combination tablet LY900010 (5 mg LY2452473 with a smaller particle size #1, d90 = 10 microns, and 5 mg tadalafil) administered orally, once.
  There was a washout period of at least 7 days between each intervention. d90 is a measurement of the distribution of particle widths such that 90% of the particles have a diameter less than the specified value.
Period: First Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: First Washout Period of 1 Week
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Second Washout Period of 1 Week
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Third Washout Period of 1 Week
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All randomized participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24
Race, Customized [Count of Participants; unit: Participants]
  Black or African American | 4
  White | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve From Time Zero to Infinity [AUC(0-∞)] of LY2452473
Time Frame: Predose up to 96 hours postdose for each of the 4 treatment periods
Population: Entire study population: All randomized participants.
Measure: Mean (Standard Deviation); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- 5 mg LY2452473 and 5 mg Tadalafil: Participants who were administered a 5-milligram (mg) LY2452473 capsule and 5-mg tadalafil tablet during any study period.
- LY900010 (Particle Size #1): Participants who were administered a single combination tablet LY900010 (containing 5 mg LY2452473 with a smaller particle size #1, d90 = 10 microns, and 5 mg tadalafil) during any study period.
- LY900010 (Particle Size #2): Participants who were administered a single combination tablet LY900010 (containing 5 mg LY2452473 with an intermediate particle size #2, d90 = 25 microns, and 5 mg tadalafil) during any study period.
- LY900010 (Particle Size #3): Participants who were administered a single combination tablet LY900010 (containing 5 mg LY2452473 with a larger particle size #3, d90 = 40 microns, and 5 mg tadalafil) during any study period.
Arm/Group | 5 mg LY2452473 and 5 mg Tadalafil | LY900010 (Particle Size #1) | LY900010 (Particle Size #2) | LY900010 (Particle Size #3)
Number analyzed (Participants) | 24 | 24 | 24 | 24
nanograms*hours per milliliter (ng*h/mL) | 514 (152) | 495 (159) | 453 (123) | 463 (140)
Statistical Analysis 1: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs LY900010 (Particle Size #1); Test type: Non-Inferiority or Equivalence — AUC(0-∞) was log-transformed and analyzed using a linear mixed effects model with fixed factor for formulation, sequence, and period, and random factor for participant; Geometric Least Squares (LS) Mean Ratio = 0.96, 90% CI 2-sided [0.91 to 1.01] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs LY900010 (Particle Size #2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric LS Mean Ratio = 0.89, 90% CI 2-sided [0.85 to 0.93] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 3: Comparison: LY900010 (Particle Size #1) vs LY900010 (Particle Size #2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric LS Mean Ratio = 0.93, 90% CI 2-sided [0.88 to 0.97] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 4: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs LY900010 (Particle Size #3); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric LS Mean Ratio = 0.90, 90% CI 2-sided [0.86 to 0.95] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 5: Comparison: LY900010 (Particle Size #1) vs LY900010 (Particle Size #3); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric LS Mean Ratio = 0.94, 90% CI 2-sided [0.90 to 0.99] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 6: Comparison: LY900010 (Particle Size #2) vs LY900010 (Particle Size #3); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric LS Mean Ratio = 1.02, 90% CI 2-sided [0.97 to 1.07] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor

2. Primary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of LY2452473
Time Frame: Predose up to 96 hours postdose for each of the 4 treatment periods
Population: Entire study population: All randomized participants.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- LY900010 (Particle Size #2): Participants who were administered a single combination tablet LY900010 (containing 5 mg LY2452473 with an intermediate particle size# 2, d90 = 25 microns, and 5 mg tadalafil) during any study period.
Arm/Group | 5 mg LY2452473 and 5 mg Tadalafil | LY900010 (Particle Size #1) | LY900010 (Particle Size #2) | LY900010 (Particle Size #3)
Number analyzed (Participants) | 24 | 24 | 24 | 24
nanograms per milliliter (ng/mL) | 32.5 (8.16) | 27.1 (6.62) | 25.6 (7.41) | 24.7 (5.66)
Statistical Analysis 1: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs LY900010 (Particle Size #1); Test type: Non-Inferiority or Equivalence — Cmax was log-transformed and analyzed using a linear mixed effects model with fixed factor for formulation, sequence, and period, and random factor for participant; Geometric LS Mean Ratio = 0.84, 90% CI 2-sided [0.77 to 0.91] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs LY900010 (Particle Size #2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric LS Mean Ratio = 0.78, 90% CI 2-sided [0.71 to 0.85] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 3: Comparison: LY900010 (Particle Size #1) vs LY900010 (Particle Size #2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric LS Mean Ratio = 0.93, 90% CI 2-sided [0.85 to 1.01] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 4: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs LY900010 (Particle Size #3); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric LS Mean Ratio = 0.77, 90% CI 2-sided [0.70 to 0.84] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 5: Comparison: LY900010 (Particle Size #1) vs LY900010 (Particle Size #3); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric LS Mean Ratio = 0.91, 90% CI 2-sided [0.84 to 1.00] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 6: Comparison: LY900010 (Particle Size #2) vs LY900010 (Particle Size #3); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Geometric LS Mean Ratio = 0.99, 90% CI 2-sided [0.91 to 1.08] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor

3. Secondary Outcome: Pharmacokinetics: AUC(0-∞) of Tadalafil
Time Frame: Predose up to 96 hours postdose for each of the 4 treatment periods
Population: Entire study population: All randomized participants.
Measure: Mean (Standard Deviation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | 5 mg LY2452473 and 5 mg Tadalafil | LY900010 (Particle Size #1) | LY900010 (Particle Size #2) | LY900010 (Particle Size #3)
Number analyzed (Participants) | 24 | 24 | 24 | 24
nanograms*hours per milliliter (ng*h/mL) | 2410 (893) | 2400 (1070) | 2240 (676) | 2290 (825)
Statistical Analysis 1: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs LY900010 (Particle Size #1); Test type: Superiority or Other; Geometric LS Mean Ratio = 0.99, 90% CI 2-sided [0.93 to 1.05]
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs LY900010 (Particle Size #2); Test type: Superiority or Other; Geometric LS Mean Ratio = 0.94, 90% CI 2-sided [0.89 to 1.00]
Statistical Analysis 3: Comparison: LY900010 (Particle Size #1) vs LY900010 (Particle Size #2); Test type: Superiority or Other; Geometric LS Mean Ratio = 0.96, 90% CI 2-sided [0.90 to 1.02]
Statistical Analysis 4: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs LY900010 (Particle Size #3); Test type: Superiority or Other; Geometric LS Mean Ratio = 0.96, 90% CI 2-sided [0.90 to 1.02]
Statistical Analysis 5: Comparison: LY900010 (Particle Size #1) vs LY900010 (Particle Size #3); Test type: Superiority or Other; Geometric LS Mean Ratio = 0.97, 90% CI 2-sided [0.91 to 1.03]
Statistical Analysis 6: Comparison: LY900010 (Particle Size #2) vs LY900010 (Particle Size #3); Test type: Superiority or Other; Geometric LS Mean Ratio = 1.01, 90% CI 2-sided [0.95 to 1.08]

4. Secondary Outcome: Pharmacokinetics: Cmax of Tadalafil
Time Frame: Predose up to 96 hours postdose for each of the 4 treatment periods
Population: Entire study population: All randomized participants.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- LY900010 (Particle Size #1): Participants who were administered a single combination tablet LY900010 (5 mg LY2452473 with a smaller particle size #1, d90 = 10 micron, and 5 mg tadalafil) during any study period.
- LY900010 (Particle Size #2): Participants who were administered a single combination tablet LY900010 (5 mg LY2452473 with an intermediate particle size #2, d90 = 25 micron, and 5 mg tadalafil) during any study period.
- LY900010 (Particle Size #3): Participants who were administered a single combination tablet LY900010 (5 mg LY2452473 with a larger particle size #3, d90 = 40 micron, and 5 mg tadalafil) during any study period.
Arm/Group | 5 mg LY2452473 and 5 mg Tadalafil | LY900010 (Particle Size #1) | LY900010 (Particle Size #2) | LY900010 (Particle Size #3)
Number analyzed (Participants) | 24 | 24 | 24 | 24
nanograms per milliliter (ng/mL) | 102 (31.2) | 74.4 (28.0) | 72.4 (19.0) | 70.0 (17.5)
Statistical Analysis 1: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs LY900010 (Particle Size #1); Test type: Superiority or Other; Geometric LS Mean Ratio = 0.72, 90% CI 2-sided [0.68 to 0.77] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 2: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs LY900010 (Particle Size #2); Test type: Superiority or Other; Geometric LS Mean Ratio = 0.71, 90% CI 2-sided [0.66 to 0.76] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 3: Comparison: LY900010 (Particle Size #1) vs LY900010 (Particle Size #2); Test type: Superiority or Other; Geometric LS Mean Ratio = 0.98, 90% CI 2-sided [0.92 to 1.05] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 4: Comparison: 5 mg LY2452473 and 5 mg Tadalafil vs LY900010 (Particle Size #3); Test type: Superiority or Other; Geometric LS Mean Ratio = 0.69, 90% CI 2-sided [0.65 to 0.74] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 5: Comparison: LY900010 (Particle Size #1) vs LY900010 (Particle Size #3); Test type: Superiority or Other; Geometric LS Mean Ratio = 0.96, 90% CI 2-sided [0.90 to 1.02] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor
Statistical Analysis 6: Comparison: LY900010 (Particle Size #2) vs LY900010 (Particle Size #3); Test type: Superiority or Other; Geometric LS Mean Ratio = 0.98, 90% CI 2-sided [0.91 to 1.04] — Formulation, sequence, and period were included in the model as fixed effects, and participant as a random factor

ADVERSE EVENTS:
Groups:
- 5 mg LY2452473 and 5 mg Tadalafil: Participants who were administered a 5-mg LY2452473 capsule and 5-mg tadalafil tablet during any study period.
Arm/Group | 5 mg LY2452473 and 5 mg Tadalafil | LY900010 (Particle Size #1) | LY900010 (Particle Size #2) | LY900010 (Particle Size #3)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 3/24 | 7/24 | 5/24 | 3/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg LY2452473 and 5 mg Tadalafil (N=24) | LY900010 (Particle Size #1) (N=24) | LY900010 (Particle Size #2) (N=24) | LY900010 (Particle Size #3) (N=24)
Scleral hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensation of pressure (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site swelling (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 5 (5) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Penis disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days